CLINICAL TRIAL: NCT07276230
Title: Quality of Life Assessment of Caregivers of Patients With Multiple Myeloma Participating in a Therapeutic Education Program and Receiving a Supportive Care Needs Evaluation
Brief Title: Quality of Life Assessment of Caregivers of Patients With Multiple Myeloma
Acronym: ENTRAIDANT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP250083
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Caregivers of Patients With Multiple Myeloma
Keywords: caregivers; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Caregivers

STUDY DESIGN:
Intervention Model Description: Caregivers of patients followed for multiple myeloma during first-line therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregivers (Experimental): Therapeutic Education and Needs Assessment Program for Caregivers of Patients with Multiple Myeloma
  Interventions: Other: Therapeutic Education and Needs Assessment Program for Caregivers

INTERVENTIONS:
Other: Therapeutic Education and Needs Assessment Program for Caregivers — Participation in a weekly therapeutic education group for 4 weeks.

SUMMARY:
The diagnosis and treatment of multiple myeloma affect not only the patient but also their family and caregivers. Advances in therapy have transformed the follow-up of patients treated for multiple myeloma. The involvement of informal caregivers has become increasingly essential to ensure adequate home-based care, as most treatments are now delivered on an outpatient basis. Literature reviews suggest that caregivers of cancer patients often face unmet supportive care needs, which in turn negatively impact their quality of life.

DETAILED DESCRIPTION:
By improving the quality of life of caregivers, the intervention can help prevent cascading effects such as a deterioration in the quality of life of the care recipient, thereby reducing the overall burden on healthcare systems. In addition, therapeutic education is an ongoing process aimed at helping patients and/or caregivers acquire or maintain the skills they need to best manage their lives with a chronic condition.

Study procedures :

1. During the hematology consultation, the study will be presented to the caregiver identified by the patient (between Day -7 and Day 0). After receiving full oral and written information, the caregiver's free, written, and informed consent will be obtained prior to participation.
2. After providing written informed consent to participate in the study, the caregiver will attend an individual interview at Day 0 with a nurse to complete a Shared Educational Assessment .The caregiver will then independently complete a self-administered questionnaire assessing quality of life using the CarGOQoL (CareGiver Oncology Quality of Life).

   The Shared Educational Assessment is a discussion between the healthcare professional and the caregiver focusing on the skills to be acquired or strengthened in order to improve health and quality of life. It enables exploration and assessment of the caregiver's needs and resources in terms of :
   * Acquisition of knowledge;
   * Acquisition or reinforcement of self-care and coping skills, while recognizing and valuing the caregiver's own self learning efforts.
3. The group of caregivers thus constituted will attend four therapeutic education workshops. Each workshop will last approximately 1 hour and 30 minutes. Caregivers will attend two half-day sessions, participating in two workshops per session (Week 1: Workshops 1 & 2; Week 2: Workshops 3 & 4).

   The topics addressed in the workshops are as follows:
   * Workshop 1: Understanding the disease
   * Workshop 2: Identifying abnormalities in biological tests and adapting the appropriate response
   * Workshop 3: Understanding treatments and their adverse effects
   * Workshop 4: Expressing personal experiences and feelings caregivers' satisfaction with each workshop will be assessed at the end of every session
4. At the end of the program (three months after inclusion), the caregiver will attend a follow-up consultation with the nurse to evaluate skill acquisition and will independently complete the same quality of life questionnaire (CarGOQoL) that was administered prior to the program
5. At six months, a new assessment of quality of life will be conducted using the CarGOQoL questionnaire during a telephone interview with a member of the investigative team

The questionnaire will be available in paper format, and the responses will be entered into an electronic case report form (e-CRF) using the CleanWeb system. The data will be analyzed by the Clinical Research Unit (URC).

ELIGIBILITY:
Inclusion Criteria:

Caregiver :

* Designated by a patient followed for multiple myeloma during first-line treatment
* Providing weekly assistance to the patient (e.g., shopping, housekeeping, management of daily living activities, healthcare or hygiene support, etc.)
* Aged 18 years or older
* Fluent in French
* Affiliated with or benefiting from a social security system (excluding state medical aid - AME)
* Able to provide free, written, and informed consent

Exclusion Criteria:

Caregiver :

* Not designated by the patient as the primary caregiver
* Currently being treated for an acute medical condition
* Refusal of the caregiver to participate in the study
* Under legal protection (guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of a needs assessment approach through participation in a therapeutic education program on improving the quality of life of caregivers of patients with multiple myeloma. | 3 months
  Change in caregivers' CarGOQoL (CareGiver Oncology Quality of Life) scores between baseline and 3 months. The higher the score, the better the quality of life.

SECONDARY OUTCOMES:
Caregivers' adherence to the therapeutic education program for caregivers of patients with multiple myeloma | 3 months
  Proportion of caregivers who completed the entire therapeutic education program
Changes in caregivers' specific skills after participation in the program (self-care and coping skills) | 6 months
  Assessment of self-care and coping skills using a four-level competency acquisition scale: acquired, not acquired, introduced, and reinforcement session required
Caregivers' satisfaction with participation in the workshops | 2 weeks
  Caregivers' satisfaction measured using a Visual Analogue Scale (VAS) ranging from 1 to 10. The higher the score, the greater the satisfaction.
The long-term effectiveness of this approach on caregivers' quality of life. | 6 months
  Change in caregivers' CarGOQoL (CareGiver Oncology Quality of Life) scores between baseline and 6 months. The higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Anne LE BORGNE, Mrs, Principal Investigator — Hospital Pitié Salpêtrière - Assistance Publique Hôpitaux de Paris
Locations (1):
- Hématologie clinique - Pitié-Salpêtrière Hospital (APHP), Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.